CLINICAL TRIAL: NCT00939159
Title: Phase II Study of LBH589 for Patients With Low or Intermediate-1 Risk Myelodysplastic Syndrome
Brief Title: Study of LBH589 for Patients With Low or Intermediate-1 Risk Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0713
Record Dates: First submitted 2009-07-10; First posted 2009-07-14 (Estimated); Results first posted 2015-06-18 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: Myelodysplastic Syndrome
Keywords: Low or Intermediate-1 Risk Myelodysplastic Syndrome; MDS; Cancer; LBH589
MeSH Terms: conditions — Myelodysplastic Syndromes; Neoplasms | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LBH589 (Experimental): LBH589 20 mg capsules by mouth 3 times a week for 3 weeks in a 28-day cycle.
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589 — 20 mg capsules by mouth 3 times a week for 3 weeks in a 28-day cycle.

SUMMARY:
The goal of this clinical research study is to learn if LBH589 can help to control lower-risk (low or intermediate-1 risk) MDS. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
Study Drug:

LBH589 is a drug that may slow down the growth of cancer cells or kill cancer cells by blocking certain enzymes (proteins produced by cells).

Study Drug Administration:

If you are found to be eligible to take part in this study, you will take LBH589 capsules by mouth 3 times a week for 3 weeks (for example on Days 1, 3, 5, 8, 10,12, 15, 17, and 19) then 1 week of rest of each 28-day study "cycle."

You should take LBH589 at the same time each morning. Each dose of LBH589 should be taken with 1 cup (8 ounces) of water.

You should swallow the capsules whole and not chew them. You must not eat grapefruit and Seville (sour) oranges or drink their juices during your entire participation on the study.

If you vomit while taking LBH589, then you should wait until your next scheduled dose to take another capsule. If you forget to take your capsules in the morning, you can take them up to 12 hours after the usual time you take it. After 12 hours, do not take LBH589 that day. Instead, wait until your next scheduled dose. Do not make up missed doses.

Call your study doctor or study staff as soon as possible if you have any unusual symptoms. Do not wait until your next visit to tell your doctor about your symptoms. If you have side effects at your assigned dose level, then your dose may be lowered. You may also have to stop taking LBH589 for a short period, and the side effect(s) will be watched by your doctor until they resolve.

Take the drug just as the doctor tells you. Do not miss any capsules. You will be asked to return all study drug in the bottles provided, whether your take all the capsules or not. Empty bottles should also be brought back to the clinic. Capsules should not be transferred between bottles at any time.

At each visit, you must tell the study staff about any other drugs you are taking during the study. This includes prescription drugs, over-the-counter drugs, and vitamins. Your study doctor will tell you if you need to stop taking any of these drugs.

Study Visits:

At least every week during Cycle 1 and every cycle after that, you will have the following tests and procedures performed:

* Blood (about 1 tablespoon) will be drawn for routine tests
* You will have a physical exam, including measurement of your vital signs.

On Day 21 (+/- 7 days) of Cycle 1, you will have a bone marrow biopsy/aspirate to check the status of the disease.

On Days 1 and 5 of Cycle 1, and Days 5 and 22 of Cycles 2 and beyond, you will have ECGs. If your doctor thinks it is necessary, you may have ECGs more often.

On Day 1 of Cycle 2 and beyond you will have EKG prior to taking the study medication.

Length of Study:

You may continue taking the study drug for up to 24 months. You will be taken off study if intolerable side effects occur or the disease gets worse.

End of Study Visit:

When you stop taking LBH589, you will have the following tests and procedures performed:

* Blood (about 1 tablespoon) will be drawn for routine tests
* You will have a bone marrow aspiration and biopsy to check the status of the disease.
* You will have a physical exam, including measurement of your vital signs.
* You will have a performance status evaluation.
* You will have an ECG.

This is an investigational study. LBH589 is not FDA approved or commercially available. At this time, LBH589 is only being used for research.

Up to 40 participants will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with intermediate-1 risk MDS or transfusion dependent low risk MDS by the IPSS classification. Patient must have one or more cytopenia as defined by IPSS (Cytopenias are defined as an absolute neutrophil count < 1800 K/uL; or hemoglobin < 10 g/dl or platelets < 10^5 K/uL).
2. Signed informed consent indicating that patients are aware of the investigational nature of this study prior to participation in the study and any related procedures being performed.
3. Age >/= 18 years old
4. Prior therapy with growth factor support, lenalidomide, 5-azacytidine, decitabine or other investigational agents is allowed if last dose was given more than 14 days prior to first dose of LBH 589.
5. Previously untreated patients are eligible for this study.
6. Patients must meet the following laboratory criteria: AST/SGOT and ALT/SGPT </= 2.5 x upper limit of normal (ULN) or </= 5.0 x ULN if the transaminase elevation is due to leukemic involvement; Serum bilirubin </= 1.5 x ULN; Serum creatinine </= 1.5 x ULN or 24-hour creatinine clearance >/= 50 ml/min; Serum potassium >/= lower limit of normal (LLN); Serum phosphorous >/= LLN; Serum total calcium (corrected for serum albumin) or serum ionized calcium >/= LLN; Serum magnesium >/= LLN; TSH and free T4 within normal limits (WNL) (patients may be on thyroid hormone replacement)
7. Baseline MUGA or ECHO must demonstrate LVEF >/= the lower limit of the institutional normal of 50%.
8. ECOG Performance Status of </= 2
9. Women of childbearing potential (WOCBP) defined as not post-menopausal for 12 months or no previous surgical sterilization must have a negative serum pregnancy test within 72 hours of the first administration of oral LBH589.
10. Male patients who agree to use a condom during sexual contact with a female of child bearing potential.
11. Patients with a heart rate >/= 50 beats per minute with or without a pacemaker.

Exclusion Criteria:

1. Prior treatment with an HDAC inhibitor for MDS or any other malignancy.
2. Patients currently treated with valproic acid for neurological or other conditions who can not be changed to another therapy.
3. Impaired cardiac function including any one of the following: Screening ECG with QTc > 450 msec confirmed by central laboratory prior to enrollment in study; Pts with congenital long QT syndrome; History of sustained ventricular tachycardia; History of ventricular fibrillation or torsades de pointes; Pts with myocardial infarction or unstable angina within 6 mo. of study entry; Congestive heart failure; Right bundle branch block with left anterior hemiblock (bifascicular block)
4. Concomitant use of drugs with a risk of causing torsades de pointes. A wash-out period of at least 72 hours is required. Patients using medications that have a relative risk of prolonging the QT interval or inducing torsades de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug.
5. Concomitant use of CYP3A4 inhibitors. A wash-out period of at least 72 hours is required.
6. Patients with unresolved diarrhea greater than CTCAE grade 1
7. Patients who have undergone major surgery less than 4 weeks prior to screening visit or who have not recovered from side effects of such therapy.
8. Patients who have received chemotherapy, any investigational drug or undergone major surgery within 3 weeks prior to starting study drug or who have not recovered from side effects of such therapy (CTCAE Grade 1), with the exception of nitrosoureas, which should be discontinued at least six weeks before enrollment.
9. Concomitant use of any anti-cancer therapy or radiation therapy.
10. Patients with a history of another primary malignancy within 5 years other than curatively treated CIS of the cervix, or basal or squamous cell carcinoma of the skin
11. Patients with known positivity for human immunodeficiency virus (HIV) ) or hepatitis C.
12. Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent
13. Female patients who are pregnant or breastfeeding.
14. Uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen.
15. Impairment of GI function or GI disease that may significantly alter the absorption of LBH589
16. Peripheral neuropathy greater than CTCAE grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-08; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Study Chair — UT MD Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Dimicoli S, Jabbour E, Borthakur G, Kadia T, Estrov Z, Yang H, Kelly M, Pierce S, Kantarjian H, Garcia-Manero G. Phase II study of the histone deacetylase inhibitor panobinostat (LBH589) in patients with low or intermediate-1 risk myelodysplastic syndrome. Am J Hematol. 2012 Jan;87(1):127-9. doi: 10.1002/ajh.22198. Epub 2011 Nov 10. PMID 22072492
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: August 05, 2009 to March 10, 2011. All recruitment done at The University of Texas (UT) MD Anderson Cancer Center.
Pre-assignment Details: Of the seventeen (17) participants enrolled, four were excluded prior to receiving treatment on the study.
Period: Overall Study
Arm/Group | LBH589
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LBH589
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 70 [47 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Based on the Hematologic Improvement
Description: Overall response rate defined by International Working Group (IWG) response criteria in myelodysplasia. Hematologic Improvement (HI) responses, at least 9 weeks: Erythroid response (pretreatment, <11 g/dL): Hgb increase by 1.5 g/dL; Relevant reduction units of Red blood cell (RBC) transfusions by absolute number at least 4 RBC transfusions/8 week compared with pretreatment transfusion number in previous 8 weeks; Only RBC transfusions for Hgb of 9.0 g/dL pretreatment count in RBC transfusion response evaluation; Platelet response (pretreatment,<100x10^9/L): If starting with >20x10^9/L platelets:
  absolute increase 30x10^9/L, Increase from baseline <20 x10^9/L to >20x10^9/L and by =/> 100%; Neutrophil response (pretreatment, <1.0x10^9/L): =/> 100% increase & absolute increase >0.5x10^9/L; Progression or relapse after HI: At least 1 of the following: =/>50% decrement from max response levels in granulocytes or platelets; Reduction in Hgb by 1.5 g/dL; or Transfusion dependence .
Time Frame: Assessment with 28-day cycle until response, then every 3 cycles as needed, for up to 24 months
Population: Of the seventeen participants registered, four were not treated making thirteen evaluable for response.
Measure: Number; unit: Percentage of Participants
Arm/Group | LBH589
Number analyzed (Participants) | 13
Percentage of Participants | 8

ADVERSE EVENTS:
Time Frame: Adverse event collected for eligible participants each three week treatment cycle. Overall study period: August 06, 2009 to March 17, 2011.
Arm/Group | LBH589
Serious Adverse Events (participants affected / at risk) | 4/13
Other Adverse Events (participants affected / at risk) | 3/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LBH589 (N=13)
Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated to study drug
QTc Prolongation (Cardiac disorders) | 1 (1)
Cholecystitis (Infections and infestations) | 1 (1) — Unrelated to study drug
Death/Disease Progression (General disorders) | 1 (1) — Unrelated to study drug
Confusion (Nervous system disorders) | 1 (1) — Unrelated to study drug
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LBH589 (N=13)
Fatigue (General disorders) | 2 (2)
Decreased appetite (Gastrointestinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 2

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes